CLINICAL TRIAL: NCT02576743
Title: Pushing Spatiotemporal Limits for 4D Flow MRI and Dynamic MRA in the Brain at Ultra-High Field
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1508M77106
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: Stroke; AVM; Aneurysm
MeSH Terms: conditions — Stroke; Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy subjects: Subjects with no contraindications to magnetic resonance imaging will undergo 4D flow MRI scanning. 7 Tesla MRI
  Interventions: Device: 7 Tesla MRI
- Patients: Patients with an unruptured brain aneurysm or an unruptured arteriovenous malformation (AVM) with no contraindications to magnetic resonance imaging will undergo 4D flow MRI scanning 7 Tesla MRI
  Interventions: Device: 7 Tesla MRI

INTERVENTIONS:
Device: 7 Tesla MRI — MR imaging using a 7 Tesla MR system.

SUMMARY:
This study aims at investigating the blood hemodynamics with high spatiotemporal resolution in patients with brain aneurysms and AVMs as well as in healthy controls. Parameters such as peak blood velocity, wall shear stress and other derived parameters will be obtained from 4D flow MRI data acquired at ultra-high field strength (7 Tesla).

DETAILED DESCRIPTION:
The hemodynamic factors responsible for hemorrhagic stroke, resulting in wide variations in the clinical management of underlying vascular lesions, especially when they are found in asymptomatic individuals or individuals with symptoms not related to the disease. Therefore, there is an urgent need for the development of reliable biomarkers based on hemodynamic parameters, which can then enable improvements in risk assessment in patients presenting with these lesions. This need can be met by non-invasive Magnetic Resonance Imaging (MRI) techniques that provide information on high resolution vascular anatomy, visualization of cerebral hemodynamics and quantitative information about blood velocity. However, such techniques as presently employed at 1.5 or 3 Tesla are limited by spatial resolution and prolonged data acquisition times.

The primary goal of this proposal is to overcome these current limitations by exploiting Ultra-High Fields (UHF, i.e. ≥ 7 Tesla (7T)) to attain significantly higher spatial resolution, faster acquisitions and increased lesion conspicuity utilizing

* Qualitative exploration of intracranial blood hemodynamics,
* Quantitative imaging of the spatiotemporally resolved blood velocity vector,
* Derivation of hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects / Patients between 18 and 75

Exclusion Criteria:

* Any kind of ferromagnetic implants.
* MR-unsafe non-ferromagnetic implants.
* Cardiac pacemakers.
* A history of shrapnel or shot gun injury.
* A body mass index > 40.
* Severe claustrophobia.
* Tattoos in the head/neck area or permanent makeup.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients, age 18-75 years;
  * Patients with previously un-ruptured AVMs, who have had a catheter-guided DSA for evaluation of the AVM; any Spetzler-Martin grade; patients with one or more un-ruptured AVMs regardless of symptoms
  * Patients with non-symptomatic patients; one or more un-ruptured conservatively managed aneurysms, all aneurysm sizes and shapes (fusiform, saccular, sessile).
  Subjects:
  - healthy subjects between 18 and 75 years.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Brain Flow Dynamics | 2 years
  Altered brain flow hemodynamics in patients with aneurysms and AVMs compared to normal subjects

CONTACTS AND LOCATIONS:
Overall Officials: Bharathi Jagadeesan, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States